CLINICAL TRIAL: NCT00962312
Title: A Phase II Study of Lapatinib and Capecitabine in the Treatment of Metastatic Pancreatic Cancer.
Brief Title: Lapatinib Ditosylate and Capecitabine in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-39 ICORG; ICORG-08-39; EUDRACT-2008-006907-22; EU-20933
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2012-10

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Lapatinib

ARMS (1):
- Capecitabine and Lapatinib (Experimental)
  Interventions: Drug: capecitabine; Drug: lapatinib ditosylate

INTERVENTIONS:
Drug: capecitabine
Drug: lapatinib ditosylate

SUMMARY:
RATIONALE: Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib ditosylate together with capecitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving lapatinib ditosylate together with capecitabine works in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of lapatinib ditosylate and capecitabine as first-line therapy, in terms of overall survival, in patients with metastatic pancreatic cancer.

Secondary

* To evaluate the progression-free survival of patients treated with this regimen.
* To evaluate the overall response rate (complete and partial responses) in patients treated with this regimen.
* To evaluate the clinical benefit (complete response, partial response, or stable disease for ≥ 6 months) of this regimen in these patients.
* To evaluate the qualitative and quantitative toxicity associated with this regimen in these patients.
* To determine the intra-tumoral expression of ErbB1 (EGFR) and ErbB2 (HER2/neu) in these patients.
* To seek pilot information on the intra-tumoral expression of markers of tumor resistance and sensitivity to treatment, including resistance drug pump expression and growth factor receptor expression.
* To collect pre- and post-treatment serum samples from these patients for proteomic analyses to elucidate if any serum cancer marker profiles can be detected.

OUTLINE: This is a multicenter study.

Patients receive oral lapatinib ditosylate once daily on days 1-21 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas
* Measurable or non-measurable disease

  * Measurable disease is defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No known brain metastases or leptomeningeal disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Albumin ≥ 2.5 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN) (2.5 times ULN if Gilbert's syndrome is present)
* AST and ALT ≤ 3 times ULN (5 times ULN if documented liver metastases are present)
* Creatinine < 1.5 times ULN
* Cardiac ejection fraction normal by ECHO or MUGA scan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow and retain oral medication
* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, requirement for IV alimentation, or uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* No active hepatic or biliary disease, except for Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment
* No active cardiac disease within the past 6 months, including any of the following:

  * Uncontrolled angina
  * Clinically significant arrhythmia, except for asymptomatic atrial fibrillation requiring anticoagulation
  * Myocardial infarction
  * Uncontrolled or symptomatic congestive heart failure
  * Any other cardiac condition that, in the opinion of the treating physician, would make this study unreasonably hazardous for the patient
* No concurrent uncontrolled illness including, but not limited to, ongoing or active infection or psychiatric illness/social situation that would limit compliance with study requirements
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to lapatinib ditosylate or any of its excipients, capecitabine, or fluorouracil
* No known dihydropyrimidine dehydrogenase (DPD) deficiency
* No other malignancy within the past 5 years except for completely resected nonmelanoma skin cancer or successfully treated in situ carcinoma

PRIOR CONCURRENT THERAPY:

* Recovered from prior radiotherapy or surgery
* No prior surgical procedures affecting absorption
* No prior EGFR- or ErbB2-targeting therapies
* No prior capecitabine
* No prior chemotherapy for locally advanced or metastatic pancreatic cancer
* At least 3 months since prior adjuvant chemotherapy

  * Prior fluorouracil allowed as a radiosensitizer only
* More than 30 days (or 5 half-lives) since prior investigational drugs
* No concurrent radiotherapy or surgery for metastatic cancer
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent CYP3A4 inducers or inhibitors
* No other concurrent investigational agents or anticancer therapy (e.g., cytotoxic or biologic therapy)
* No concurrent herbal (alternative) medicines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
6-month survival rate | 6 months

SECONDARY OUTCOMES:
Progression-free survival | 6 months
  Progression-free survival (PFS) will be measured as the number of days between patient's enrolment and his or her date of progression of disease. Patients who are still living six months after the last patient has been enrolled will be censored for the analyses, using the number of days between enrolment and the date of last follow-up. Disease progression will be determined according to definitions established in the modified response evaluation criteria in solid tumours (RECIST) (refer to Appendix G). For patients with non-measureable tumours disease progression will be determined by the treating physician in consultation with the Chief investigator for the study.
Overall response rate | up to 6 months
  The overall response rate will be an aggregation of the complete responses and partial responses. For patients to be given the status of complete response or partial response a confirmatory disease assessment should be performed no less than four weeks after the criteria for response are first met.
Clinical benefit | 6 months
  A patient will be regarded as' having experienced clinical benefit if they have shown a complete response, a partial response, or stable disease for at least six months.
Safety and tolerability | Throughout course of study
Tumour biomarker analysis | Currently ongoing
  Characterising the patient population by determination of intra-tumoural expression of ErbB1 (EGFR) and ErbB2 (Her2/neu).Seeking pilot information as to the intra-tumoural expression of markers of tumour resistance and sensitivity to treatment. Proteomic analysis of serum samples for potential markers.

CONTACTS AND LOCATIONS:
Overall Officials: Ray McDermott, MD, Principal Investigator — Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital
Locations (9):
- Ireland (9):
  - Cork University Hospital, Cork
  - Mercy University Hospital, Cork
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University College Hospital, Galway